CLINICAL TRIAL: NCT06429449
Title: Mitoxantrone for Venetoclax Resistant Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-0178.cc; NCI-2024-04761 (Other: CTRP)
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Leukemia; Myeloid Leukemia; Monocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Monocytic, Acute | interventions — venetoclax; Azacitidine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will be a conventional 3+3 dose-escalation study to determine maximum tolerated (MTD) or recommended dose of mitoxantrone when used with venetoclax+azacitidine.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Mitoxantrone
- Cohort 2 (Experimental): After establishing the MTD of mitoxantrone, an expansion cohort will open. 10 subjects refractory to first-line therapy w/venetoclax+HMA, or respond then relapse after first-line therapy w/venetoclax+HMA, will enroll in the study & receive a subsequent cycle of venetoclax+azacitidine at the dose & schedule being administered per the standard of care, w/the determined MTD/recommended dose of IV mitoxantrone given days 1-4. Day 28 +/- 7 days of this cycle, a bone marrow biopsy will be repeated. In the absence of a ≥50% blast reduction from baseline, the subject will discontinue the study. If a CR, CRi, MLFS or blast reduction from baseline of ≥50% occurs, the subject can continue sequential cycles of venetoclax+azacitidine at the dose & schedule being administered per the standard of care, with the MTD/recommended dose of mitoxantrone on days 1-4, up to 3 cycles. No subject will receive >3 cycles of mitoxantrone.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Mitoxantrone
- Cohort 3 (Experimental): Subjects in a morph remission w/ MRD+ after ≤3 cycles of soc ven+HMA will enroll & receive mitox on days 1-4 at dose tbd that is below the MTD from cohort 1, concurrently w/ven+aza, at the dose & schedule being soc admin, over a 28-day cycle. A BMBX w/ MRD assessment will be done day 28. If MRD- occurs, subseq treatment cycles will continue to admin ven+aza, at the dose & schedule being soc admin, w/ the tbd dose of mitox on days 1-4, for max of 3 cycles. If MRD- does not occur, the next cycle may escalate the mitox dose to a level tbd & not exceeding the MTD, w/ ven+aza at the dose & schedule being soc admin. If MRD- occurs, subseq treatment cycles will continue to admin ven+aza, at the dose & schedule being soc admin, with the tbd dose of IV mitox on days 1-4, for a max of 3 cycles. If MRD- does not occur, the next cycle may escalate the mitox to a level tbd & not exceeding the MTD, w/ ven+aza at the dose & schedule being admin per the soc. Subjects will not receive >3 cycles.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Mitoxantrone
- Cohort 4 (Experimental): Subjects in a morphologic remission w/ MRD+ after >3 cyc of soc ven/HMA will enroll 28-50 days after the previous ven/HMA cyc. Subjects will receive mitox IV days 1-4 at a dose tbd below the MTD from cohort 1; on day 14, the subject will start ven+aza at the dose & schedule per the soc. On day 42, a BMBX, w/ MRD assessment, will be repeated. If MRD- occurs, subseq cyc will cont to admin ven+aza, at the dose & schedule per the soc, with the tbd dose of IV mitox on days 1-4, for a max of 3 cyc of mitox. If MRD- does not occur, the next cyc will retain the same schedule & may escalate the mitox to a dose level tbd & not exceeding the MTD. If MRD- occurs, 1 add'l cyc of mitox at this dose, w/ ven+aza at the dose & schedule per the soc, will be given. If MRD- does not occur, the next cyc will retain the same schedule & may escalate the mitox to a level tbd & not exceeding the MTD.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Venetoclax — Venetoclax attaches to a protein called Bcl-2. This protein is present in high amounts in CLL cancer cells, where it helps the cells survive for longer in the body and makes them resistant to cancer medicines. By attaching to Bcl-2 and blocking its actions, venetoclax causes the death of cancer cells and thereby slows down progression of the disease.
  Other Names: Venclexta; Venclyxto
Drug: Azacitidine — An analog of the pyrimidine nucleoside cytidine, has effects on cell differentiation, gene expression, and deoxyribonucleic acid (DNA) synthesis and metabolism, and causes cytotoxicity.
  Other Names: Onureg; Vidaza
Drug: Mitoxantrone — Mitoxantrone Injection, USP (concentrate) is a synthetic antineoplastic anthracenedione for intravenous use.
  Other Names: Novantrone

SUMMARY:
This is an open label, phase 1 study for AML subjects with relapsed or refractory disease or subjects in morphologic remission with MRD+ after first line therapy with venetoclax+HMA. A preliminary dose-finding cohort will be followed by 3 expansion cohorts.

DETAILED DESCRIPTION:
This is an open label, phase 1 study for AML subjects with relapsed or refractory disease or subjects in morphologic remission with MRD+ after first line therapy with venetoclax+HMA. A preliminary dose-finding cohort will be followed by 3 expansion cohorts.

Cohort 1 will be a conventional 3+3 dose-escalation study to determine maximum tolerated (MTD) or recommended dose of mitoxantrone when used with venetoclax+azacitidine. Subjects who are refractory to first-line therapy with venetoclax+HMA, or who respond and then relapse after first line therapy with venetoclax+HMA, will enroll in the study and receive a subsequent cycle of venetoclax+azacitidine at the dose and schedule being administered per the standard of care, along with a starting dose of 2mg/m2 of mitoxantrone administered IV on days 1-4. Depending on the absence or frequency of dose-limiting toxicities, additional patients will be enrolled at the appropriate dose levels, increasing by 2mg/m2 per cycle, per the 3+3 design until the MTD or a dose of 10mg/m2 of mitoxantrone is reached. The dose escalation phase will conclude when the MTD is determined; if the MTD is not reached, a recommendation for a dose of mitoxantrone in combination with venetoclax+azacitidine will be made based on toxicity and efficacy data.

After the establishment of the MTD or recommended dose of mitoxantrone, an expansion cohort (cohort 2) will open. 10 subjects who are refractory to first-line therapy with venetoclax+HMA, or who respond and then relapse after first line therapy with venetoclax+HMA, will enroll in the study and receive a subsequent cycle of venetoclax+azacitidine at the dose and schedule being administered per the standard of care, with the determined MTD/recommended dose of IV mitoxantrone given on days 1-4. On day 28 +/- 7 days of this cycle, a bone marrow biopsy will be repeated. In the absence of a ≥50% blast reduction from baseline, the subject will discontinue the study. If a CR, CRi, MLFS or blast reduction from baseline of ≥50% occurs, the subject can continue sequential cycles of venetoclax+azacitidine at the dose and schedule being administered per the standard of care, with the MTD/recommended dose of mitoxantrone on days 1-4, for up to 3 total cycles. No subject will receive >3 cycles of mitoxantrone. After mitoxantrone cycles have been completed, subjects will receive a bone marrow biopsy after the third cycle, and then continue bone marrow biopsies with MRD assessments every 6 months, until disease progression or the administration of any therapy other than venetoclax+azacitidine, at which time the subject will be discontinued from the study.

In cohort 3, subjects who are in a morphologic remission with MRD+ after ≤3 cycles of standard of care venetoclax+HMA will enroll and receive mitoxantrone on days 1-4 at a dose to-be-determined that is below the MTD from cohort 1, concurrently with venetoclax+azacitidine, at the dose and schedule being administered per the standard of care, over a 28-day treatment cycle. A bone marrow biopsy with MRD assessment will be performed on day 28 +/- 7 days. If MRD conversion to negative occurs, subsequent treatment cycles will continue to administer venetoclax+azacitidine, at the dose and schedule being administered per the standard of care, with the to-be-determined dose of mitoxantrone on days 1-4, for a maximum of three total cycles of mitoxantrone. If MRD conversion to negative does not occur, the next cycle may escalate the mitoxantrone dose to a level to-be-determined and not exceeding the MTD, with venetoclax+azacitidine at the dose and schedule being administered per the standard of care. If MRD conversion to negative occurs, subsequent treatment cycles will continue to administer venetoclax+azacitidine, at the dose and schedule being administered per the standard of care, with the to-be-determined dose of IV mitoxantrone on days 1-4, for a maximum of three total cycles of mitoxantrone. If MRD conversion to negative does not occur, the next cycle may escalate the mitoxantrone to a level to-be-determined and not exceeding the MTD, with venetoclax+azacitidine at the dose and schedule being administered per the standard of care. Subjects will not receive >3 cycles of mitoxantrone. After mitoxantrone cycles have been completed, subjects will continue bone marrow biopsies with MRD assessments every 6 months, until disease progression or the administration of any therapy other than venetoclax+azacitidine, at which time the subject will be discontinued from the study.

In cohort 4, subjects who are in a morphologic remission with MRD+ after >3 cycles of standard of care venetoclax/HMA will enroll 28-50 days after the start of the previous venetoclax/HMA cycle. They will receive mitoxantrone IV on days 1-4 at a dose to-be-determined that is below the MTD from cohort 1; on day 14, the subject will start venetoclax+azacitidine at the dose and schedule being administered per the standard of care. On day 42 +/- 7 days, a bone marrow biopsy, with MRD assessment, will be repeated. If MRD conversion to negative occurs, subsequent treatment cycles will continue to administer venetoclax+azacitidine, at the dose and schedule being administered per the standard of care, with the to-be-determined dose of IV mitoxantrone on days 1-4, for a maximum of three total cycles of mitoxantrone. If MRD conversion to negative does not occur, the next cycle will retain the same schedule, and may escalate the mitoxantrone to a dose level to-be-determined and not exceeding the MTD. If MRD conversion to negative occurs, one additional cycle of mitoxantrone at this dose, with venetoclax+azacitidine at the dose and schedule being administered per the standard of care, will be given. If MRD conversion to negative does not occur, the next cycle will retain the same schedule, and may escalate the mitoxantrone to a level to-be-determined and not exceeding the MTD. No subject will receive >3 cycles of mitoxantrone. After mitoxantrone cycles have been completed, subjects will continue bone marrow biopsies with MRD assessments every 6 months, until disease progression or the administration of any therapy other than venetoclax+azacitidine, at which time the subject will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have confirmation of non-APL AML by WHO criteria and have been treated with first-line venetoclax/HMA (azacitidine or decitabine).
2. Subject must have relapsed disease per IWG criteria or disease refractory to first line venetoclax/HMA defined by less than a PR response after ≥ 1 complete cycle of venetoclax/HMA.
3. Subject must have either measurable residual disease (MRD+), as measured by FDA-approved flow cytometric test performed by Hematologics (cohort 3 and 4) or relapsed/refractory disease (cohort 1 and 2).
4. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status of ≤ 2.
5. Subject must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 60 mL/min, calculated using the formula CKD-EPI Creatinine Equation
6. Subject must have adequate heart function as measured by left ventricular ejection fraction (LVEF) >50%, assessed by multigated acquisition (MUGA) or echocardiogram (ECHO) within 1 month prior to study day 1
7. Subject must have adequate liver function as demonstrated by:

   1. aspartate aminotransferase (AST) ≤ 3.0 × ULN*
   2. alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   3. bilirubin ≤ 1.5 × ULN, unless due to Gilbert's syndrome*

      * Unless considered due to leukemic organ involvement
8. Non-sterile male subjects must use contraceptive methods with partner(s) at least prior to beginning study drug administration and continuing up to 90 days after the last dose of study drug. No contraception is required if male subjects are surgically sterile (vasectomy with medical assessment confirming surgical success) or if the male subject has a female partner who is postmenopausal or permanently sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Female subjects must be either:

   1. Postmenopausal; defined as Age > 60 years with no menses for 12 or more months without an alternative medical cause; OR
   2. Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy); OR
   3. If subject is of childbearing potential, use of contraception is required while on study treatment and for 6 months after the last dose.
10. Subject must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any research directed procedures.

Exclusion Criteria:

1. Subject has known active CNS involvement from AML.
2. Subject has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

   1. Significant active cardiac disease within the previous 6 months including: New York Heart Association heart failure > class 2, unstable angina, or myocardial infarction.
   2. Renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia.
3. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration. This includes history of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis), celiac disease (e.g.

   sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity.
4. Subject exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial or fungal). Uncontrolled is defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment.
5. Subject has a history of other malignancies prior to study entry, with the exception of:

   1. Adequately treated in situ carcinoma of the breast or cervix uteri
   2. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
   3. Prostate cancer not requiring therapy beyond hormonal therapy
   4. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
6. Subject has a white blood cell count > 25 × 109/L. Note: hydroxyurea or apheresis are permitted to meet this criterion (cohort 3 only).
7. Pregnant or breast-feeding females.
8. Known or suspected hypersensitivity to azacitidine or mannitol.
9. Any prior exposure to an anthracycline or anthracenedione

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Reassessment at end of each cycle (28 days) until MTD reached, up to 5 cycles total if needed
  Cohort 1: Determine the maximum tolerated (MTD) and/or recommended phase 2 dose (RP2D) of mitoxantrone in combination with venetoclax+azacitidine.
Overall response rate | Baseline to End of Treatment (up to 1 year)
  Cohort 2: Overall response rate (CR+CRi+PR+MLFS) after treatment with mitoxantrone and venetoclax+azacitidine
Number of grade 4 or 5 adverse events | Baseline to End of Treatment (up to 1 year)
  Cohorts 3 and 4: determine the safety of mitoxantrone in combination or in sequence with standard of care venetoclax+azacitidine

SECONDARY OUTCOMES:
Survival data | Through study completion, up to 5 years
  All cohorts: Relapse free survival, remission duration, overall survival and adverse events by grade and attribution
Number of conversions from MRD+ to MRD- | After each cycle of treatment (28 days), up to 3 cycles total
  Cohorts 3 and 4: Determine the rate of conversion from MRD+ to MRD- after treatment with mitoxantrone.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kent, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No